CLINICAL TRIAL: NCT02850445
Title: Effects of Integrated Treatment for Chinese Patients With Schizophrenia: 1-year Follow-up
Brief Title: Trial and Follow-up of the Efficacy of Two-stage Integrated Treatment for Chinese Schizophrenia Inpatients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Responsible Party: Principal Investigator, Shenglin She, Clinical Professor, Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Huiai 2014Y2-00105
Record Dates: First submitted 2016-07-14; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Cognitive Behavioral Therapy; Rehabilitation; Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Integrated Treatment (Experimental)
  Interventions: Drug: Olanzapine; Other: Cognitive behavior therapy; Other: Rehabilitation treatment; Other: Case management
- antipsychotic medication alone treatment (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — All patients with schizophrenia were under medication treatment at the baseline. Individualized plan of antipsychotic medication for the patients were determined by psychiatrist who were blind to the group allocation. Medications could be changed at any time during the course of the study if the change was clinically warranted, the drug can also be any other antipsychotic medication.
Other: Cognitive behavior therapy — Patients with schizophrenia allocated to the Integrated Treatment(IT) group received Cognitive behavioral therapy.
  Arms: Integrated Treatment
Other: Rehabilitation treatment — Rehabilitation treatment include three modules: medication management, symptom management, and social kill training. Patients with schizophrenia allocated to the Integrated Treatment(IT) group received Rehabilitation treatment therapy.
  Arms: Integrated Treatment
Other: Case management — Patients with schizophrenia allocated to the Integrated Treatment(IT) group received Case management.
  Arms: Integrated Treatment

SUMMARY:
Regular psychosocial intervention combined with antipsychotic drugs, compared with usual medication alone treatments, can reduce psychiatric symptoms and improve quality of life in patients with schizophrenia. However, it's expensive, time-consuming, and sometimes inconvenient for patients and their family members in developing areas where the number of well-trained therapist remains limited in local psychiatric settings. The investigators aimed to establish an efficient model of integrated treatment (IT) for patients with schizophrenia. The procedure contains two stages: a centralized treatment during hospitalization and the following consolidation treatments with long intervals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with the Structured Clinical Interview for DSM-IV (SCID-DSM-IV) (First et al., 1996), were recruited from inpatient psychiatric ward. Patients with diagnoses of schizoaffective or other psychotic disorders were not included.
* Additional inclusion criteria for participants were aged between 18 and 50 years with education of more than 9 years, and
* PANSS (Positive and Negative Syndrome Scale) total scores of more than 60.

Exclusion Criteria:

* Diagnosed with a serious and unstable medical condition including abuse and/or dependence of alcohol and/or drugs;
* Pregnant or breastfeeding;
* Under a treatment of clozapine with a dose of more than 200 mg/day,
* Had a treatment of the electroconvulsive therapy (ECT) or modified electroconvulsive therapy within 6 months(MECT) within the past six months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Medication nonadherence was assessed in two groups after 12-month follow-up. | One year follow-up
  Medication non-adherence was defined as a failure to take medication for one week or longer
Rehospitalization rate was assessed in two groups after 12-month follow-up. | One year follow-up
Rate of Relapse was assessed in two groups after 12-month follow-up. | One year follow-up

SECONDARY OUTCOMES:
Improvement of symptoms in each group was assessed by the change of PANSS(Positive and Negative Syndrome Scale) total scale score. | One year follow-up
  Time course and treatment differences for changes in the PANSS( Positive and Negative Syndrome Scale) was analyzed using Mixed-Effects Model for Repeated-Measures analyses (MMRM).
Improvement of symptoms in each group was assessed by the change of CGI( Clinical Global Impressions) scale score. | One year follow-up
  Time course and treatment differences for changes in the CGI( Clinical Global Impressions) was analyzed using Mixed-Effects Model for Repeated-Measures analyses (MMRM).
Social functioning in each group was assessed by the change of PSP(Personal and Social Performance)scale score. | One year follow-up
  Time course and treatment differences for changes in the PSP(Personal and Social Performance) were analyzed using Mixed-Effects Model for Repeated-Measures analyses (MMRM).

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou psychitric hosptial, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] She S, Deng Y, Chen Y, Wu C, Yi W, Lu X, Chen X, Li J, Li R, Zhang J, Xiao D, Wu H, Ning Y, Zheng Y. Two-stage integrated care versus antipsychotic medication alone on outcomes of schizophrenia: One-year randomized controlled trial and follow-up. Psychiatry Res. 2017 Aug;254:164-172. doi: 10.1016/j.psychres.2017.04.054. Epub 2017 Apr 25. PMID 28463714